CLINICAL TRIAL: NCT06341517
Title: Brain Circuitry Therapeutics for Schizophrenia - A Cross-species Longitudinal Randomized Controlled Clinical Study to Treat Negative Symptoms of Schizophrenia Using Non-invasive Stimulation of the Cerebellum
Brief Title: Brain Circuitry Therapeutics for Schizophrenia
Acronym: ATHENA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indrit Begue (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Indrit Begue, Assistant Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC-ID:2023-D0117
Record Dates: First submitted 2023-12-04; First posted 2024-04-02 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects, care providers, investigators and outcome assessors will all be blinded as to the randomization sequence, and thus will be blinded as to sham vs active TMS status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active intermittent theta burst stimulation (iTBS) to the cerebellum at 80% of active motor threshold.
  Interventions: Device: iTBS
- Placebo (Placebo Comparator): Sham intermittent theta burst stimulation (iTBS) to the cerebellum
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — Intermittent Theta Burst Stimulation (iTBS) pattern consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses for up to 8 sessions daily for 5 days

SUMMARY:
This project is a double blind randomized clinical trials that examines the efficacy of cerebellar non invasive stimulation for apathy improvement in patients with schizophrenia

DETAILED DESCRIPTION:
This double-blind RCT aims to explore the efficacy of intensiveTranscranial Magnetic Stimulation (TMS) in schizophrenia spectrum disorders. Previous studies in various disorders suggest that intensive TMS is efficacious and safe.

Participants will undergo neuronavigated intermittent theta burst TMS, targeted to individual network targets, at an accelerated protocol (multiple sessions a day), The primary goal is to determine the efficacy of this protocol in alleviating negative symptoms of schizophrenia.

Additionally, the study will measure the impact of accelerated TMS on a range of clinical and cognitive outcomes, along with neuroimaging markers indicative of symptom response.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Capable of giving informed consent as evaluated by the treating psychiatrist
  * Informed Consent signed by the subject
  * Patients aged 18 - 65 years diagnosed with a schizophrenia spectrum disorder (including schizophrenia, schizoaffective or non-organic psychosis, psychotic disorder NOS) according to DSM-5 criteria
  * Clinically stable condition judged by their treating psychiatrist
  * Background antipsychotic medication treatments have remained unchanged for at least 4 weeks
  * No hospitalization in acute psychiatry ward at least 3 months prior to study entry

Specific exclusion criteria related to psychopathology

* Comorbid and clinically active current major depressive episode determined by the treating psychiatrist.
* Active psychotic symptoms. In particular, patients that at Baseline have a PANSS scores of more than 4 in any of the following PANSS items: delusions, suspiciousness/persecution and hallucinatory behaviour will be considered not stable enough to participate.
* Significant extrapyramidal side-effects quantified by total score of mSAS > 12.
* Increased sedation due to use of medication (slowing, drowsiness, slurred speech etc.)
* Active daily use of substances (i.e. cocaine), including for therapeutically medical purposes (e.g., methadone substitution)

Exclusion criteria related to MRI or TMS

* History of fainting spells of unknown or undetermined aetiology that might constitute seizures
* History of multiple seizures or diagnosis of epilepsy
* Any progressive (e.g., neurodegenerative) neurological disorder such as multiple sclerosis or Parkinson's disease
* Chronic uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* Metallic objects/implants (excluding dental fillings) unless cleared to be MRI compatible (i.e. MRI compatible joint replacement)
* Any implants controlled by physiological signs in/near the head

  * Pacemaker
  * Implanted medication pump
  * Vagal nerve stimulator
  * Deep brain stimulator or TENS unit
  * Ventriculo-peritoneal shunt
  * Cochlear implant
* Impaired ability to sense heat/pain, open wounds etc.
* Increased intracranial pressure
* Intracranial lesion, from a known genetic disorder or from acquired neurologic disease (e.g. stroke, tumor, cerebral palsy, severe head injury, or significant dysmorphology).
* History of head injury resulting in prolonged loss of consciousness (>15minutes) or neurological sequelae
* Ongoing pregnancy and breastfeeding. All participants capable of becoming pregnant will be required to have active contraception; any participant who is pregnant or breastfeeding will not be enrolled in the study.

Other exclusion criteria

* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, cancer, pulmonary decompensation etc.)
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, intellectual retardation, dementia, etc. of the subject
* Having legal obligation for psychiatric treatment.
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation.
* Previous enrolment into the current investigation
* Enrolment of the PI, his/her family members, employees and other dependent persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Brief Negative Symptoms Scale - apathy subscale (BNSS-Apathy) at follow-up (FU) at T3. The primary endpoint will be assessed at baseline and all follow-up visits at week 1, 6 and 12. | at 12 weeks
  This outcome measure focuses on the evaluation of changes in apathy symptoms in participants, utilizing the apathy subscale of the Brief Negative Symptoms Scale (BNSS-Apathy).
  Apathy symptoms will be assessed at baseline (pre-intervention) and subsequently at follow-up visits scheduled at weeks 1, 6, and 12 post-intervention. The primary endpoint of this measure is the change in BNSS-Apathy scores from baseline to each follow-up point, aiming to capture the trajectory of symptom changes across the study period.
  The BNSS-Apathy subscale score, derived from specific item responses, provides a quantitative measure of apathy severity, allowing for statistical analysis of symptom changes over time. Higher scores reflect greater severity of symptoms. Maximum score of BNSS-Apathy subscale score is 42 (severe apathy), minimum score is 0.

SECONDARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) positive and negative subscores at follow-up | at 1 week
  This outcome measure focuses on the evaluation of apathy and psychosis symptoms
Positive and Negative Symptoms Scale (PANSS) positive and negative subscores at follow-up | at 6 weeks
  This outcome measure focuses on the evaluation of apathy and psychosis symptoms
Positive and Negative Symptoms Scale (PANSS) positive and negative subscores at follow-up | at 12 weeks
  This outcome measure focuses on the evaluation of apathy and psychosis symptoms
Self reported Negative Scale SNS scores and its sub-scales at follow-up | at 1 week
  This outcome measure focuses on the self-reported evaluation of apathy
Self reported Negative Scale SNS scores and its sub-scales at follow-up | at 6 weeks
  This outcome measure focuses on the self-reported evaluation of apathy
Self reported Negative Scale SNS scores and its sub-scales at follow-up | at 12 weeks
  This outcome measure focuses on the self-reported evaluation of apathy
Brief neurocognitive assessment (BNA) scores at follow-up | at 6 weeks
  This outcome measure focuses on the evaluation of cognitive function
Auditory Hallucinations Rating Scale (AHRS) scores at follow-up | at 6 weeks
  This outcome measure focuses on the evaluation of auditory hallucinations
Calgary Depression Scale (CDSS) scores at follow-up | at 6 weeks
  This outcome measure focuses on the evaluation of depression symptoms
Young Mania Rating Scale (YMRS) scores at follow-up | at 6 weeks
  This outcome measure focuses on the evaluation of mania symptoms
Personal and social performance scale (PSP) scores at follow-up | at 12 weeks
  This outcome measure focuses on the evaluation of psychosocial functioning
Deep-phenotyping outcome - sEBR (spontaneous eye blink) | at 6 weeks
  This outcome measure focuses on the evaluation of sEBR
Deep-phenotyping outcome - facial expressions | at 6 weeks
  This outcome measure focuses on the evaluation of facial expressions
Deep-phenotyping outcome - accelerometer | at 6 weeks
  This outcome measure focuses on the evaluation of accelerometry
Cerebellar-cortical functional connectivity | at 1 week
  This outcome measure focuses on cerebellar-cortical functional connectivity
Cerebellar-cortical structural connectivity | at 6 weeks
  This outcome measure focuses on cerebellar-cortical structural connectivity
Cerebellar-cortical structural connectivity | at 12 weeks
  This outcome measure focuses on cerebellar-cortical structural connectivity

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Campus Biotech, Geneva
  - Indrit Bègue, Geneva

IPD SHARING:
Plan to Share IPD: Undecided